CLINICAL TRIAL: NCT03563885
Title: Effect of Bariatric Surgery on Tissue-specific Glucose Uptake
Brief Title: Glucose Uptake in Metabolic Tissues After Bariatric Surgery
Acronym: GU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Financial and Method issues suggesting that study is not feasible.
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 304180015
Record Dates: First submitted 2018-06-08; First posted 2018-06-20 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Obesity; Insulin Resistance
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RYGB or SG (Experimental): Baseline testing followed by subject's already scheduled RYGB or SG surgery, and then post-testing.
  Interventions: Procedure: bariatric surgery
- Lean (No Intervention): Lean control subjects doing baseline testing only.

INTERVENTIONS:
Procedure: bariatric surgery — subjects already scheduled Roux-en-Y gastric bypass (RYGB) or sleeve gastrectomy (SG) surgery
  Arms: RYGB or SG

SUMMARY:
The goal of this study is to provide a comprehensive evaluation of whole-body and tissue-specific glucose metabolism after consuming a mixed meal in lean people and people with obesity, before and after 20-35% weight loss induced by Roux-en-Y gastric bypass or sleeve gastrectomy surgery.

DETAILED DESCRIPTION:
Obesity is associated with an impairment in postprandial glucose disposal, which is an important risk factor for type 2 diabetes (T2D). Weight loss improves postprandial glycemic control. The difficulty in achieving successful weight loss by using lifestyle therapy (diet and physical activity) has led to an increased interest in bariatric surgery, which is the most effective available weight loss therapy. Moreover, bariatric surgery procedures that bypass the upper gastrointestinal tract, such as Roux-en-Y gastric bypass (RYGB) and sleeve gastrectomy (SG), have profound effects on glycemic control and cause remission in a large percentage of people with T2D. However, the effect of RYGB and SG surgery on postprandial glucose disposal among key metabolic organs has not been investigated and compared. The goal of this study is to provide a comprehensive evaluation of whole-body and tissue-specific glucose metabolism after consuming a mixed meal in lean people and people with obesity, before and after 20-35% weight loss induced by RYGB or SG surgery. Glucose uptake (GU) will be assessed by using: i) a combination of oral and intravenous stable isotopically-labeled glucose tracers to assess the delivery of ingested glucose into the systemic circulation and whole-body glucose disposal rate; and ii) positron emission tomography (PET) with magnetic resonance (MR) imaging to assess muscle, subcutaneous and visceral adipose tissue, liver, small intestine, and pancreas GU.

ELIGIBILITY:
Inclusion Criteria:

* BMI 35.0-50.0 kg/m2 for obese group and 18.5-24.9 kg/m2 for the lean group
* Must be scheduled for RYGB or SG surgery

Exclusion Criteria:

* Previous bariatric surgery
* Unstable weight (>4% change during the last 2 months before entering the study)
* Significant organ system dysfunction (e.g., severe pulmonary or kidney disease)
* Cancer or cancer that has been in remission for <5 years
* Conditions that render subject unable to complete all testing procedures (e.g. metal implants that interfere with imaging procedures; coagulation disorders)
* Use of medications that are known to affect the study outcome measures or increase the risk of study procedures and that cannot be temporarily discontinued for this study
* Pregnant or lactating women
* Persons who are not able to grant voluntary informed consent
* Persons who are unable or unwilling to follow the study protocol or who, for any reason, the research team considers not an appropriate candidate for this study, including non-compliance with screening appointments or study visits

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity | An average of 6 months from baseline testing to 20-35% weight loss
  Insulin sensitivity will be assessed by positron emission topography & magnetic resonance imaging before and after bariatric surgery

CONTACTS AND LOCATIONS:
Overall Officials: George Schweitzer, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Center for Human Nutrition, St Louis, Missouri, United States